CLINICAL TRIAL: NCT02551536
Title: Comparison of Efficacy, Safety and Cost Effectiveness of Montelukast and Levocetirizine Versus Montelukast and Fexofenadine in Patients of Allergic Rhinitis: a Randomized, Double-blind Clinical Trial
Brief Title: Montelukast and Fexofenadine Versus Montelukast and Levocetrizine Combination in Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indira Gandhi Medical College, Shimla (Other)
Responsible Party: Principal Investigator, DR.MOHINI MAHATME, ASSOCIATE PROFESSOR, Indira Gandhi Medical College, Shimla
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/425-26/13
Record Dates: First submitted 2015-08-12; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; montelukast; fexofenadine; levocetrizine
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast; fexofenadine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): FDC tablet of montelukast 10 mg and levocetrizine 5 mg was given once daily for 4 weeks
  Interventions: Drug: Montelukast; Drug: Levocetrizine
- Group B (Experimental): FDC tablet of montelukast 10 mg and fexofenadine 120 mg was given once daily for 4 weeks
  Interventions: Drug: Montelukast; Drug: Fexofenadine

INTERVENTIONS:
Drug: Montelukast
Drug: Fexofenadine — group B received FDC tablet of montelukast 10mg and fexofenadine 120 mg O.D
  Arms: Group B
Drug: Levocetrizine — group A recieved FDC tablet of montelukast 10 mg and levocetrizine 5mg O.D
  Arms: Group A

SUMMARY:
Objectives: Allergic Rhinitis (AR) is a global health problem. 10-25% of population worldwide is affected by AR. Oral/intranasal H1-antihistamine, decongestants, leukotriene receptor antagonists, intranasal corticosteroids are the pillars in the management of AR.Materials and methods: Seventy patients with allergic rhinitis participated in a prospective, randomized, double-blind, parallel, active controlled, comparative 4 week trial. The patients between age group of 18-65 years of either gender having moderate-severe intermittent or mild persistent allergic rhinitis were included. The study inclusion criteria required the subjects with Total Nasal Symptom Score (TNSS) of 5 or higher. The patients were randomly divided into two treatment groups with montelukast-levocetrizine (10 mg and 5 mg) in one group and montelukast-fexofenadine (10 mg and 120 mg) in another group. TNSS parameter was the main effectiveness parameter.

DETAILED DESCRIPTION:
Allergic Rhinitis (AR) is a global health problem. It is the cause of major illness and disability worldwide. Estimates indicate that 10-25% of population worldwide is affected by AR. The main symptoms of AR include nasal congestion, rhinorrhea, itching, sneezing and non-nasal symptoms like burning, itching and watery eyes or itching ears and palate. These symptoms can have a considerable toll on patient's quality of life by interfering with cognitive and emotional functioning. The estimated annual cost attributable to AR in United States ranges from $1.4 billion to nearly $ 6 billion in direct cost annually. Today's antiallergic therapy is based on avoidance of the causative allergen, symptomatic pharmacotherapy, specific immunotherapy and education. Oral/intranasal H1-antihistaminics, decongestants, leukotrienes receptor antagonists, intranasal corticosteroids are the pillars in the management of allergic rhinitis. Second generation antihistamines have become increasingly popular because of their comparable efficacy and lower incidence of adverse effects relative to first generation counterparts. Levocetirizine, a potent second generation histamine (H1) receptor antagonist, is effective against persistent allergic rhinitis and thus improves quality of life and reduces co-morbidities and societal costs. Fexofenadine, is a selective, non sedating, second generation H1 receptor antagonist which have an additional impact on the inflammatory mediators. Monteleukast is a highly selective type I receptor antagonist of leukotriene D4. The leukotrienes modifiers have both anti-inflammatory and bronchodilator properties.

The literature search establishes that addition of an antihistamine to montelukast has added benefit. The combination therapy of montelukast with antihistamine provide enhancing and complimentary effects thereby reducing the symptoms effectively. The results with concomitant levocetirizine and montelukast treatment are better as compared to monotherapy with levocetirizine on symptoms and quality of life in allergic rhinitis. Fexofenadine along with montelukast is more effective than antihistaminic alone in control of allergic rhinitis symptoms. There is literature available for the comparisons of concomitant levocetirizine and montelukast with monotherapy or placebo and comparisons of concomitant fexofenadine and montelukast with monotherapy or placebo. But scanty data is available regarding comparisons of concomitant montelukast-levocetirizine with montelukast-fexofenadine.

ELIGIBILITY:
Inclusion Criteria:

* either gender having moderate-severe intermittent or mild persistent allergic rhinitis according to original Aria classification.
* subjects with Total Nasal Symptom Score (TNSS) of 5 or higher.
* not treated with antihistaminics in previous week.
* Patients willing to sign written informed consent
* free of any clinically significant disease
* having normal E.C.G

Exclusion Criteria:

* participation of children, pregnant female, nursing mothers,
* patients with asthma requiring chronic use of inhaled or systemic corticosteroids
* history of failure to improve symptoms with antihistaminic drug treatment in the past 4.history of allergies to study medication or tolerance to antihistamines, 5.use of study drug in the last 7 days. 6. subjects with significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric or autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 4 week
  The TNSS was obtained from the sum of all four individual symptom scores, with a total possible score ranging from 0 (no symptoms) to 12 (maximum symptom intensity).
adverse drug reaction | 4 week
  General clinical safety was monitored by vigilant follow-up of patients for the treatment of emergent adverse events if any, and recorded in the case report form

SECONDARY OUTCOMES:
cost effectiveness ratio | 4 weeks
  direct cost parameters were taken into consideration. Direct cost parameters were cost of medications used, medical procedures and hospitalization charges, if any. Cost-effectiveness ratio of both treatment groups were calculated based on formula as given below.
  Cost-effectiveness ratio = cost / outcome Outcome was measured in terms of effectiveness. TNSS parameter was the main effectiveness parameter.